CLINICAL TRIAL: NCT02594345
Title: In Vitro Study of the Effect of Exosomes Derived From Red Blood Cell Units on Platelet Function and Blood Coagulation in Healthy Volunteers' Blood
Brief Title: Effect of Exosomes Derived From Red Blood Cell Units on Platelet Function and Blood Coagulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Dr Dania Fischer, Research associate, Johann Wolfgang Goethe University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ExoRBC
Record Dates: First submitted 2015-10-30; First posted 2015-11-03 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Blood Coagulation; Platelet Function
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention group (Experimental)
  Interventions: Other: in vitro study

INTERVENTIONS:
Other: in vitro study — Exosomes will be mixed with healthy volunteers' blood in vitro

SUMMARY:
This study is designed to analyze the effect exosomes derived from red blood cell units have on blood coagulation and platelet function. It is an in vitro study using healthy volunteers' blood.

DETAILED DESCRIPTION:
The blood of 25 healthy volunteers will be exposed to exosomes derived from red blood cell units. The effects on coagulation and platelet function will be measured using thromboelastometry (ROTEM®) and FACS analysis.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* pregnancy
* drug use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
clotting time | 2 months
  measured by thromboelastometry (ROTEM® Analysis)

SECONDARY OUTCOMES:
clot formation | 1h after exposure
  measured by thromboelastometry (ROTEM® Analysis)
clot stability | 1h after exposure
  measured by thromboelastometry (ROTEM® Analysis)
clot lysis | 1h after exposure
  measured by thromboelastometry (ROTEM® Analysis)
CD62P | 3h after exposure
  FACS analysis

CONTACTS AND LOCATIONS:
Overall Officials: Dania P Fischer, M.D., Principal Investigator — Goethe University
Locations (1):
- University Hospital Frankfurt, Frankfurt am Main, Hesse, Germany